CLINICAL TRIAL: NCT06944171
Title: Investigation of the Effects of Associated Impairments in School-Age Children With Cerebral Palsy on the Child's Activity and Participation Level and on Their Families
Brief Title: Effects of Associated Impairments on Activity and Participation in Children With Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra Erdinler, Graduate Student, Hacettepe University
Other Study IDs: HU-FTR-EE-01
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
Keywords: family; comorbidity; child; intellectual disability; cerebral palsy; epilepsy; seizures; vision disorders; hearing loss; speech disorders; caregiver; quality of life; activities of daily life; social participation
MeSH Terms: conditions — Cerebral Palsy; Intellectual Disability; Epilepsy; Seizures; Vision Disorders; Hearing Loss; Speech Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- School-aged children with Cerebral Palsy: Children with cerebral palsy between the ages of 6 and 12 volunteered for the study
- Families with children with cerebral palsy: Parents of children with cerebral palsy between the ages of 6 and 12 volunteered for the study.

SUMMARY:
This study will investigate the effects of associated impairments on the activity levels and social participation of school-aged children with Cerebral Palsy (aged 6-12) and their impact on their families' quality of life and caregiving burden.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) defines a group of permanent disorders in movement and posture development, which are expressed as non-progressive disorders that occur in the developing baby brain during life in the womb or the first 3 years after birth, causing restrictions in activity and participation.

Hearing, speech, vision, cognitive, eating and swallowing problems and epilepsy primarily accompany the motor and postural control problems seen in CP. It is reported that cognitive disabilities or learning difficulties are seen in 50-75%, speech problems in 25%, hearing problems in 25%, seizures in 25-35% and visual disorders in 40-50% of individuals with CP. These primary problems, which accompany from the beginning, vary according to the clinical type and functional effect of CP and affect the severity of the existing CP clinical picture.

The International Classification of Functioning, Disability and Health (ICF) is a framework that guides the comprehensive assessment and treatment of children with CP by considering the wide range of health-related problems they face. The ICF includes four interrelated components: body structure and functions, activity and participation, and personal and environmental factors. According to the ICF, impairments are defined as significant deviations or losses in body structure and functions, while activity limitations, difficulties in activities, and participation restrictions are defined as problems in the form or scope of participation in life.

With these impairments added to the clinical picture, children with CP face significant limitations in their activity and participation levels. Therefore, it is important to define the relationship between comorbid impairments and activity and participation limitations in order to create holistic treatment goals and interventions that improve the activity and participation levels of children with CP.

According to the World Health Organization, quality of life, especially the health-related quality of life of parents of children with special needs, is a complex and comprehensive concept related to the physical health status, psychological status, independence level, social relationships, personal beliefs and environmental characteristics of the parents.

The care of children with CP is long-term and difficult. It has been reported that frequent hospital visits from the moment of diagnosis, the need for multidisciplinary therapy and the difficulty of the care process can lead to the parents not being able to spare time for themselves and their surroundings, economic difficulties and deterioration in their quality of life.

When the literature is examined, no study has been found that examines the multidimensional problems accompanying CP, especially with a sample from our country.

ELIGIBILITY:
For children:

Inclusion criteria

* Having a diagnosis of cerebral palsy
* Being between the ages of 6-12
* Having family approval for the study Exclusion criteria
* Being under the age of 6 and over the age of 12
* Parents and children who do not volunteer to participate in the study
* Not knowing Turkish

For families:

Inclusion criteria

* Having a child between the ages of 6-12 diagnosed with cerebral palsy
* Being willing to participate in the study Exclusion criteria
* Not being willing to participate in the study
* Not knowing Turkish
* Not being able to read and write

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with CPand their families who applied to Hacettepe University Faculty of Physical Therapy and Rehabilitation Cerebral Palsy and Pediatric Rehabilitation Unit and Ministry of National Education Keçiören Guidance and Research Center and agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
PEDI-CAT (Pediatric Evaluation of Disability Inventory Computer Adaptive Test) | Single assessment conducted during the initial study visit
  The PEDI-CAT measures abilities in three functional domains: Daily Activities, Mobility and Social/Cognitive. The PEDI-CAT's Responsibility domain measures the extent to which the caregiver or child takes responsibility for managing complex, multi-step life tasks.
LIFE-H 3.0 (The Assessment of life habits) | Single assessment conducted during the initial study visit
  The Assessment of life habits (LIFE-H) is a questionnaire that is used to collect information on all life habits that people carry out in their environment (home, workplace or school, neighborhood) to ensure their survival and development in society throughout their lifetime. LIFE-H uses a numerical scoring system ranging from 0 to 9. A score of 0 indicates a complete disability or impairment in participation, while a score of 9 indicates an optimal level of participation.

SECONDARY OUTCOMES:
Nottingham Health Profile | Single assessment conducted during the initial study visit
  NSP is a scale used to assess the quality of life of families with children with cerebral palsy. This profile was developed to measure the physical, emotional and social health status of individuals. The survey consists of 7 subsections and a total of 45 items. The answers to the questions are yes/no. The participant receives 0 points for each no answer and different points for each yes answer. The maximum score that can be obtained from the survey is 607. High scores indicate low quality of life, while low scores indicate high quality of life.
Impact on Family Scale (IPFAM) | Single assessment conducted during the initial study visit
  It was developed to assess the burden of the child's illness on the family for families or caregivers of disabled children. It consists of five headings: 1) Economic burden, the extent to which the illness changes the family's economic situation, 2) Social impact, the quality and amount of interaction with other people outside the immediate family, 3) Familial impact, the quality of interaction within the family unit, 4) Personal difficulty, the subjective burden experienced by the primary caregiver, 5) Coping, the strategies used by the family to cope with the child's illness or disability. A four-point Likert-type assessment is scored from "4: I completely agree" to "1: I completely disagree." A low score from the survey indicates a high level of impact on the family.

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze Kerem-Gunel, Professor, Study Director — Hacettepe University, Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation Cerebral Palsy and Pediatric Rehabilitation Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants were informed, through the written informed consent form, that all personal data collected during the study would be kept strictly confidential and used solely for research purposes. The form also explained that their identities would not be revealed in any publication or report resulting from the study.